CLINICAL TRIAL: NCT05158348
Title: A Comparative Study to Measure the Effect of Nebulized Dexmedetomidine - Lidocaine for Controlling Postoperative Pain After Tonsillectomy in Adults.
Brief Title: A Comparative Study to Measure the Effect of Nebulized Dexmedetomidine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Mohamed, Principal investigator, lecturer of anesthesia and ICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-394-2020
Record Dates: First submitted 2021-12-07; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Dexmedetomidine; Lidocaine; Tonsillectomy
Keywords: Post tonsillectomy; Pain; Dexmedetomidine; Lidocaine
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): receive intra-operative local infiltration of saline in tonsillar bed and post-operative nebulised dexametomidine and lidocaine.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Group B (Active Comparator): receive intra-operative local infiltration of saline and post-operative will receive nebulised lidocaine
  Interventions: Drug: Nebulized lidocaine
- Group C (Active Comparator): receive intra-operative local infiltration of lidocaine and post-operative nebulised saline.
  Interventions: Drug: Local infiltration of lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Group A will receive post-operative nebulised dexametomidine and lidocaine.
  Arms: Group A
Drug: Nebulized lidocaine — Group B will receive post-operative will receive nebulised lidocaine
  Arms: Group B
Drug: Local infiltration of lidocaine — group C will receive intra-operative local infiltration of lidocaine
  Arms: Group C

SUMMARY:
A comparative study to measure the effect of nebulized dexmedetomidine - lidocaine for controlling postoperative pain after tonsillectomy in adults.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common procedures in ear, nose, and throat surgery. It is usually performed as a day-stay procedure. [1] Pain is the most common reason for physician contact after discharge, indicating that post-tonsillectomy pain is intense and undertreated. [2] Patients need analgesics that are effective and can be used safely at home.

Adults have a different pattern of pain compared with children; this is related to the different indications and techniques of tonsillectomy. [3, 4] In adults, the surgery is usually performed for chronic infection with scarred tonsils that requires dissection with coagulation, thus causing intense and longer-lasting pain. [5] In children, the indication is usually hypertrophy or recurrent acute infections with smaller changes in tonsil tissues than in adults. [6] Multimodal analgesia has become the standard of care in postoperative pain management. Combinations of analgesics with different sites or modes of action are commonly used to improve analgesia and to reduce the doses of individual analgesics (especially opioids) and to reduce adverse effects.

Systematic reviews on various analgesics for post-tonsillectomy pain have been published for paediatric and adolescent patients.(7,8) Paracetamol (alone and in combination with ibuprofen)NSAIDS,dexamethasone or gabapentenoids(9) Dexmedetomidine is a highly selective adrenergic α-2 agonist that does not cause respiratory depression and can be used as a sedative for various procedures. [10,11] Recently, the use of dexmedetomidine as an additive to local anaesthetics was reported to have several advantages over conventional intravenous administration. [12,13]

Nebulized dexmedetomidine combined with other anaesthetics as a premedication for outpatient paediatric dental procedures has also been reported to provide smoother induction of general anaesthesia with a more rapid recovery and no significant side effects. [14] Nebulized dexmedetomidine-lidocaine inhalation as a premedication for flexible bronchoscopy was well tolerated during bronchoscopies performed under moderate sedation and was associated with a reduced incidence of moderate to severe coughing, a shorter recovery time and reduced vasoconstrictor consumption(15).However, there are no data regarding the use of nebulized dexmedetomidine-lidocaine for controlling postoperative pain after tonsillectomy.

Comparative study II. Study setting and location This study will be conducted at Kasr Al-Ainy tertiary Hospital, Cairo University after being approved by the anesthesia department Research committee and obtaining written informed consent of patients III. Study population 60 patients undergoing tonsillectomy operation will be enrolled in this study divided into 3 groups each of 20 patients. Group A will receive intra-operative local infiltration of saline in tonsillar bed and post-operative nebulised dexametomidine and lidocaine. Group B will receive intra-operative local infiltration of saline and post-operative will receive nebulised lidocaine and group C will receive intra-operative local infiltration of lidocaine and post-operative nebulised saline.

IV. Eligibility Criteria

1. Inclusion criteria Patients of either sex, aged between 18-50 years old, ASA physical status I, II undergoing tonsillectomy.
2. Exclusion criteria Patients were excluded if they had clinically important coronary atherosclerotic heart disease, a history of stroke or transient ischemic attack, Sinus bradycardia or heart block, coagulopathy, peritonsillar abscess, any infection at the site of injection, Known allergy to the study drugs (lidocaine, dexmedetomidine).

V. Study Procedures

1. Randomization (in RCT only) All procedures will be performed by the same team, which include an ENT surgeon using the same technique in all study groups which is dissecting the tonsils by bipolar diathermy technique and surgeon will do the infiltration technique also and a specialized anaesthesiologist for the inhalational technique ,the patients will be informed about the procedure ,technique of the intra-operative and post-operative pain control and the VAS scoring system before the operation. Randomization and drug masking will be completed by a specialist who will not be directly involved in the trials. The patients will be divided into 3 groups; Group A will receive intra-operative local infiltration of saline in tonsillar bed and post-operative nebulised dexametomidine and lidocaine. Group B will receive intra-operative local infiltration of saline and post-operative will receive nebulised lidocaine and group C will receive intra-operative local infiltration of lidocaine and post-operative nebulised saline.

Study Protocol Upon arrival to the operating room, a pulse oximetry, capnography, continuous electrocardiogram (ECG), and non-invasive blood pressure measurement device will be connected to the patient. A large bore cannula will be inserted. Pre-medications will be given; Antiemetics as metclopromide(10mg) or dexamethasone(8mg) to decrease laryngeal edema postoperatively. Anesthesia will be induced with IV Propofol, 1.5 mg/kg and IV fentanyl 1 mic/kg and atracurium 0.5 mg/kg. Patients will be intubated and ventilated with oxygen maintaining ETCO2 at 35-40 mmHg. Anesthesia will be maintained with oxygen, isoflurane and atracurium providing muscle relaxation as a maintenance.

* Group A will receive intra-operative local infiltration of saline in tonsillar bed by the surgeon and post-operative nebulised dexametomidine(0.6mic per kg) and lidocaine(1 mic per kg)by specialized anesthesiologist. Group B will receive intra-operative local infiltration of saline by the surgeon and post-operative will receive neublised lidocaine(1 mic per kg) by specialized anesthesiologist and group C will receive intra-operative local infiltration of lidocaine(1 mic per kg) in the tonsillar bed by the surgeon and post-operative nebulised saline by the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, aged between 18-30 years old, ASA physical status I, II undergoing tonsillectomy.

Exclusion Criteria:

* Patients were excluded if they had clinically important coronary atherosclerotic heart disease, a history of stroke or transient ischemic attack, Sinus bradycardia or heart block, coagulopathy, peritonsillar abscess, any infection at the site of injection, Known allergy to the study drugs (lidocaine, dexmedetomidine).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain 4 hours after tonsillectomy measured by visual analogue score | 4 hours postoperative

SECONDARY OUTCOMES:
Postoperative nausea and vomiting following tonsillectomy operation after1 hour , 2 hours and after 4 hours | 4 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dina Mohamed, Principal Investigator — Egypt Cairo university hospitals
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided